CLINICAL TRIAL: NCT03848481
Title: Cannabidivarin (CBDV) vs. Placebo in Children and Adults up to Age 30 With Prader-Willi Syndrome (PWS)
Brief Title: CBDV vs Placebo in Children and Adults up to Age 30 With Prader-Willi Syndrome (PWS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Foundation for Prader-Willi Research (Other); GW Pharmaceuticals Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-9914
Record Dates: First submitted 2019-02-19; First posted 2019-02-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Prader-Willi Syndrome
Keywords: PWS; Prader- Willi Syndrome; Irritability; CBDV; Cannabinoids
MeSH Terms: conditions — Prader-Willi Syndrome | interventions — cannabidivarin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cannabidivarin (CBDV) (Experimental): Weight-based dosing of 10 mg/kg/day of CBDV for 12 weeks
  Interventions: Drug: CBDV Compound
- Matched Placebo (Placebo Comparator): Weight-based dosing of 10 mg/kg/day of placebo for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CBDV Compound — CBDV is obtained from the Cannabis sativa L. plant and contains a negligible quantity (less than 0.2%) of THC
  Arms: Cannabidivarin (CBDV)
Drug: Placebo — Placebo oral solution contains matching excipients.
  Arms: Matched Placebo

SUMMARY:
This study aims to examine the feasibility and safety of cannabidivarin (CBDV) as a treatment for children and young adults with PWS.

DETAILED DESCRIPTION:
This clinical research trial aims to study the feasibility and safety of cannabidivarin (CBDV), in children and young adults with Prader-Willi Syndrome (PWS). CBDV has effects independent of CB1 and CB2 receptor activation and a good safety profile. This proposal addresses the Foundation for Prader Willi Research's PWS Research Plan: Program 1, Clinical Care Research: seeks to evaluate treatments that aim to reduce behavioral symptoms, such as irritability, in order to improve the quality of life of both the individual with PWS and their families. GW Pharmaceuticals will provide the CBDV drug and matching placebo.

ELIGIBILITY:
Inclusion Criteria

1. Male or Female outpatients aged 5 to 30 years.
2. Diagnosis of PWS confirmed by genetic testing and patient medical records and history.
3. Stable pharmacologic, educational, behavioral and/or dietary interventions for 4 weeks prior to the study start, and for the duration of the study.
4. Have a physical exam and laboratory results that are within the norms for PWS
5. Presence of a parent/caregiver/guardian that is able to consent for their participation and complete assessments regarding the patient's development and behavior throughout the study. Child Assent will be obtained if the subject is 7 years of age or older and has the mental capacity to understand and sign a written assent form and/or give verbal assent.
6. Score on the Clinical Global Impression Scale Severity (CGI-S) ≥ 4 (moderate severity) at baseline.
7. Score of ≥18 on the Aberrant Behavior Checklist-Irritability (ABC-I) at baseline.
8. Agree not to drive or operate machinery.

Exclusion Criteria

1. Exposure to any investigational agent in the 30 days prior to randomization.
2. Prior chronic treatment with CBD or CBDV.
3. Positive testing for THC or other drugs of abuse via urine testing at the screening visit or baseline visits upon repeat confirmation testing.
4. History of Drug Abuse Disorder including Cannabis Use Disorder
5. A primary psychiatric diagnosis other than PWS, including bipolar disorder, psychosis, schizophrenia, PTSD or MDD. These patients will be excluded due to potential confounding results.
6. A medical condition that severely impacts the subject's ability to participate in the study, interferes with the conduct of the study, confounds interpretation of study results or endangers the subject's well-being (including but not limited to hepatic or renal impairment and cardiovascular disease).
7. Known or suspected allergy to CBDV or excipients used in the formulation (i.e. sesame).
8. Clinical indications of renal, pancreatic, or hematologic dysfunction as evidenced by values above upper limits of normal for BUN/creatinine, values twice the upper limit of normal for serum lipase and amylase, platelets <80,000 /mcL, WBC<3.0 103 /mcL. or > 2 X UNL values of AST or ALT.
9. ECG abnormality at baseline screening or clinically significant postural drop in systolic blood pressure at screening. If the initial screening ECG shows a QTcB of greater than 460 msec, then 2 additional ECGs will be conducted in the same sitting, 5 minutes apart. If not recognized at screening, then a full triplicate repeat showing an average QTcB of 460 msec or less to meet all inclusion/exclusion criteria
10. Female subjects who are pregnant will be excluded from the study. If a female subject is able to become pregnant, she will be given a pregnancy test before entry into the study. Female subjects will be informed not become pregnant while taking CBDV. Female subjects must tell the investigator and consult an obstetrician or maternal-fetal specialist if they become pregnant during the study.

Ages: 5 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Aberrant Behavior Checklist-Irritability Subscale (ABC-I) | from Baseline to Week 12
  Change in the ABC-I score. The ABC-I is a well-characterized outcome that is accepted by the FDA for the purpose of labeling, and is one of the best and most validated outcome measures in the developmental disabilities. An inclusion cutoff of 18 or higher on the ABC-I at screening was chosen based on multiple medication trials with irritability as the primary target.

SECONDARY OUTCOMES:
Repetative Behavior Scale- Revised (RBS-R) | from Baseline to Week 12
  Change in RBS-R score (a 44-item self-report questionnaire that is used to measure the breadth or repetitive behaviors)
Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS) | from Baseline to Week 12
  Change in the CY-BOCS score. The CY-BOCS is 10-item clinician measure designed to assess the severity of obsessive compulsive symptoms in children and adolescents over the previous week. It consists of four primary sections including Obsessions checklist, Severity items for Obsessions, Compulsions checklist and severity items for Compulsions and a set of investigational items. Improvement on this scale was associated with improvements in caregiver quality of life in our 8-week study of intranasal oxytocin.
Hyperphagia Questionnaire for Clinical Trials (HQ-CT) | from Baseline to Week 12
  Change in HQ-CT score. The HQ-CT is a 9-item caregiver-reported measure of food-seeking behaviors that was used in the phase 3 beloranib trial.
ActiGraph GT9X-BT activity monitors | from Baseline to Week 12
  Change in Sleep Behaviors. Actigraph activity monitors are a well validated activity sleep monitoring device that has been utilized widely in clinical trials and health research, measuring sleep latency, total sleep time, and sleep efficiency.
Clinical Global Impression Scale - Improvement (CGI-I) | from Baseline to Week 12
  The CGI-I will be used as a measure of improvement and contains a 7 point scale as follows: 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, 7 = very much worse. The CGI-I is a clinician rated global measure of improvement and has been used as a measure in previous clinical psychopharmacology trials.
Caregiver Strain Questionnaire (CSQ) | from Baseline to Week 12
  The Caregiver Strain questionnaire is a 21-item self-report questionnaire that was developed to assess caregiver strain for families with a child living with an emotional or behavioral disorder.
Montefiore Einstein Rigidity Scale-Revised-PWS (MERS-R-PWS) | from Baseline to Week 12
  The Montefiore-Einstein Rigidity Scale-Revised-PWS (MERS-R-PWS) is designed to assess three domains of rigid behavior in individuals with PWS:
  1. Behavioral Rigidity (e.g., Insistence on sameness, things must be done in his/her way, etc.)
  2. Cognitive Rigidity (e.g., Special interests, inflexible adherence to rules, etc.)
  3. Protest (in response to deviation from rigidity; e.g., tantrum, irritability, arguing) The MERS-R-PWS is a clinician-rated scale and takes about 20 minutes to complete. It will be completed only for subjects who display rigid behaviors at baseline, week 4, week 8 and week 12.
Aberrant Behavior Checklist (ABC) subscales in lethargy/social withdrawal, stereotypic behavior, hyperactivity/noncompliance, and inappropriate speech | from Baseline to Week 12
  The ABC is an informative rating instrument that was empirically derived by principal component analysis to measure behavior in those with developmental disability and ASD. It contains 58 items that resolve into 5 subscales. The subscales and the respective number of items are as follows: (a) irritability - 15 items, (b) lethargy/social withdrawal - 16 items, (c) stereotypic behavior - 7 items, (d) hyperactivity/noncompliance - 16 items, and (e) inappropriate speech - 4 items. The ABC was designed to be completed by any adult who knows the patient well, such as a parent/caregiver or teacher. This instrument measures behavior on a four-point severity scale where 0 = no problem at all, 1 = behavior is a problem but in a slight degree, 2 = problem is moderately serious, and 3 = problem is severe in degree.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hollander, MD, Principal Investigator — Montefiore Medical Center/Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center, Albert Einstein College of Medicine, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication